CLINICAL TRIAL: NCT04223167
Title: Acute Effects of Energy Drink on Hemodynamic and Electrophysiologic Parameters in Habitual and Non-Habitual Caffeine Consumers
Brief Title: Energy Drink Habituation Effects on Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Mehmet Dincer Bilgin, Professor, Aydin Adnan Menderes University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017/1211
Record Dates: First submitted 2020-01-03; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
Keywords: Energy drink; heart rate variability; habituation
MeSH Terms: conditions — Substance-Related Disorders | interventions — Water

STUDY DESIGN:
Intervention Model Description: The individuals were identified by collecting the age, weight, height, BMI, caffeine and energy drink consumption habit information by applicant acceptance questionnaire. Based on the applicant acceptance questionnaire 12 subjects were low-habitual caffeine consumers with an estimated daily intake of approximately 130 mg caffeine and named as energy drink 2 (ED2) group, 12 subjects were high-habitual caffeine consumers with an estimated daily intake of approximately more than 200 mg caffeine and named as energy drink 3 (ED3) group, while 24 subjects were caffeine naive (energy drink 1 (ED1) (n=12) and Control (n=12)) .
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Energy Drink 1 (Experimental): The participants in this group are caffeine naive and consumed 473 ml Red Bull Energy Drink
  Interventions: Dietary Supplement: Red Bull Energy Drink
- Energy Drink 2 (Experimental): The participants in this group were low-habitual caffeine consumers with an estimated daily intake of approximately 130 mg caffeine and consumed 473 ml Red Bull Energy Drink
  Interventions: Dietary Supplement: Red Bull Energy Drink
- Energy Drink 3 (Experimental): The participants in this group were low-habitual caffeine consumers with an estimated daily intake of approximately more than 200 mg caffeine and consumed 473 ml Red Bull Energy Drink
  Interventions: Dietary Supplement: Red Bull Energy Drink
- Control (Placebo Comparator): The participants in this group are caffeine naive and consumed 473 ml water
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Red Bull Energy Drink — 473 ml Reb Bull Energy Drink
  Arms: Energy Drink 1; Energy Drink 2; Energy Drink 3
Dietary Supplement: Water — 473 ml Water
  Arms: Control

SUMMARY:
The consumption of energy drinks has significantly increased in recent years but their adverse effects are not yet efficiently known. The objective of the study is to determine the acute effects of energy drink on habitual and non-habitual caffeine consumers and if caffeine consumption habit causes a difference on the hemodynamic and electrophysiologic parameters.

This study was conducted on 48 students selected from Aydın Adnan Menderes University. Four main groups were determined according to the results of the application acceptance survey. Blood pressure, electrocardiogram, breath rate, haemoglobin oxygen saturation and bioelectrical impedance analysis were measured before consuming the drinks. After consuming the drinks, measurements were repeated at 30 minutes and 60 minutes. In addition to this, Participant's Situation Anxiety Scale was applied.

DETAILED DESCRIPTION:
In this study, it is aimed to determine the acute effects of energy drink on habitual and non-habitual caffeine consumers and if caffeine consumption habit causes a difference on the hemodynamic and electrophysiologic parameters. In this respect, the complicated human body's reactions to these beverages will be examined in more detail.

Materials and methods Participants Forty eight participants (16 female, 32 male) aged 18-24 were selected from the students which are in the first year of various faculties of Aydın Adnan Menderes University. The individuals were identified by collecting the age, weight, height, BMI, caffeine and energy drink consumption habit information by applicant acceptance questionnaire. According to the results of applicant acceptance questionnaire, those with a body mass index greater than 30 kg/m2, a systemic disease, current alcoholism and smokers were not included in the study. Also, the participants who has previous adverse reactions to energy drinks were excluded to prevent undesired reactions associated with this condition. Based on the applicant acceptance questionnaire 12 subjects were low-habitual caffeine consumers with an estimated daily intake of approximately 130 mg caffeine and named as energy drink 2 (ED2) group, 12 subjects were high-habitual caffeine consumers with an estimated daily intake of approximately more than 200 mg caffeine and named as energy drink 3 (ED3) group, while 24 subjects were caffeine naive (energy drink 1 (ED1) (n=12) and Control (n=12)) . This study conforms to the Declaration of Helsinki and was approved by the Institutional Medical Ethics Committee of Adnan Menderes University (Protocol number: 2017/1211).

Experimental protocol All experiments were performed in a quiet and isolated room from external factors with room temperature of about 20°C and relative humidity between %40 and 60. All participants were advised to avoid alcohol and caffeine containing foods for at least 72 h prior to the test and to come with an overnight (12 h) fasting.

Blood pressure, electrocardiogram, breath rate, haemoglobin oxygen saturation (HOS) and BIA measurements were performed from the participants before the consumption of drinks. After the measurements ED1, ED2 and ED3 groups consumed 473 ml of Red Bull energy drink containing 151.36 mg caffeine and control group consumed the same amount of water within 5 minutes. The measurements were performed again in 30 minutes and 60 minutes. Also, state-trait anxiety inventory test (STAI) was used to assess the physiological stress of the participants.

Blood Pressure Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured indirectly by using a stethoscope (Littman Classic II, Saint Paul, USA) and aneroid sphygmomanometer (Welch Allyn Tycos, New York, USA) on each participant left arm in sitting position.

Electrocardiography (ECG) After a 5 min resting in the sitting position ECG recordings were obtained from all the individuals for 5 min in rest. Disposable Ag-AgCl electrodes were placed following the Einthoven triangle configuration. ECG measurement was performed with sampling frequency 200 Hz using ECG100C unit and BIOPAC Acqknowledge acquisition software (Biopac System Inc., Santa Barbara, CA) connected to a personal computer. PR interval, QRS complex and QTc interval values were determined from ECG recordings of the participants. QTc was calculated by Bazett's formula (QTc=QT/RR). Their normal range values are 120-200 ms, normal<140 ms and normal < 400 ms, respectively.

For acquiring the heart rate variability (HRV) time series, Pan and Thompkins algorithm was used. R peaks were detected and R-R intervals are defined. The time duration between two consecutive R peaks is termed as RR interval (tRR). The sample size of the HRV time series is 400. The heart rate (HR) is determined as:

HR=60/t_RR State-trait Anxiety Inventory (STAI) It is a test developed to determine the psychological stress during the study. STAI is defined as state and trait anxiety scale. This test is composed of two parts (40 questions). State Anxiety scale consisting of the first 20 questions was used to obtain information about the acute anxiety state of participants at the time of the study. Each question is evaluated using an ordinal scale (not at all=1, somewhat=2, moderately=3, very much=4). The total score is obtained as the sum of each answer value and gives information about the anxiety state of the participant. A total score of 50 or more is considered as positive pathological anxiety.

Haemoglobin Oxygen Saturation (HOS) HOS was measured by using a fingertip pulse oximeter on the second left finger for 1 min.

Breath Rate Breath rate measurements were taken from the participants by counting the breaths for one minute with the use of a stethoscope (Littman Classic II, Saint Paul, USA).

Bioelectrical Impedance Analysis (BIA) BIA measurements were taken by using In Body 720 before the consumption of the drinks and at 60th minute after the consumption. Each participant was asked to stand on the body composition analyzer after undressing their clothes. In Body 720 has an eight-point tactile electrode system that separately measures the impedance of the arms, trunk and legs. It measures directly the amount of the intracellular water (ICW), extracellular water (ECW), body fat percentage (PBF), body mass index (BMI) and body metabolism rate (BMR).

Statistical analysis Statistical analysis of the data was performed by using SPSS Statistics for Windows, Version 14.0. (SPSS Inc., Chicago, Illinois, USA). For comparing the groups first of all Shapiro-Wilk (SW) normality test was applied to determine the normality of the distribution. If the result of (SW) normality test was bigger than 0.05 the data were normally distributed and were analysed by using one-way analysis of variance (ANOVA) with Bonferroni post-test but if the result was less than 0.05 the data were not normally distributed and were analysed by using Kruskal-Wallis non-parametric test. Repeated ANOVA test was used for the comparison of different measurement time data of the same group. Descriptive statistics were presented as mean ± standard error of the mean (SEM). A p-value of less than 0.05 was considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between ages 18-24 years

Exclusion Criteria:

* body mass index greater than 30 kg/m2
* a systemic disease
* current alcoholism
* smokers
* the participants who has previous adverse reactions to energy drinks

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure from baseline | At baseline and 60 minutes post energy drink and placebo consumption
Change in heart rate from baseline | At baseline and 60 minutes post energy drink and placebo consumption

SECONDARY OUTCOMES:
Change in QTc interval from baseline | At baseline and 60 minutes post energy drink and placebo consumption

CONTACTS AND LOCATIONS:
Overall Officials: Serife G Caliskan, PhD., Study Director — Aydin Adnan Menderes University
Locations (1):
- Aydin Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caliskan SG, Kilic MA, Bilgin MD. Acute effects of energy drink on hemodynamic and electrophysiologic parameters in habitual and non-habitual caffeine consumers. Clin Nutr ESPEN. 2021 Apr;42:333-338. doi: 10.1016/j.clnesp.2021.01.011. Epub 2021 Feb 4. PMID 33745602